CLINICAL TRIAL: NCT05865418
Title: Feasibility and Response of a Novel Training on Dynamic Balance and Physical Activity in Adolescents With Cerebral Palsy and Spina Bifida.
Brief Title: A New Training to Enhance Physical Activity in Adolescents With Cerebral Palsy
Acronym: FOLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harshvardhan Singh, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 300011118; C-PROGRESS (Other Grant/Funding Number: C-PROGRESS); SHP RESEARCH AWARD (Other Grant/Funding Number: University of Alabama at Birmingham)
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy; Muscle Disorder; Physical Disability; Posture Disorders in Children; Spina Bifida
MeSH Terms: conditions — Cerebral Palsy; Muscular Diseases; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Adolescents with cerebral palsy will be randomly assigned to two unique exercise regimen and no exercise/standard-of-care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Loaded high intensity circuit training (Experimental): These participants will be familiarized to all the exercises. All exercises will have 3 sets, and the participants will be asked to perform as many repetitions as they can in 30s for each set. They will have 30 seconds to rest between sets (if they want more rest, we can let them more time but not exceed 60 seconds to limit the total amount of time for completing the exercise protocol) and 90 seconds to rest between exercises. Training sessions will occur twice per week with at least 24 hours between sessions. From the week 2-5 of the intervention, the participants will perform the exercises with an adjustable weight vest starting with 2.5% to finally reaching 10% of their body weight.
  Interventions: Other: Loaded high intensity training
- High Intensity Training (Active Comparator): These participants will be familiarized to all the exercises. All exercises will have 3 sets, and the participants will be asked to perform as many repetitions as they can in 30s for each set. They will have 30 seconds to rest between sets (if they want more rest, we can let them more time but not exceed 60 seconds to limit the total amount of time for completing the exercise protocol) and 90 seconds to rest between exercises. Training sessions will occur twice per week with at least 24 hours between sessions.
  Interventions: Other: High intensity circuit training (HICT)
- Control (No Intervention): They will continue their standard-of-care plan and will not involve in any new structured exercise program for 6 weeks.

INTERVENTIONS:
Other: Loaded high intensity training — Participants will be familiarized to all the exercises. All exercises will have 3 sets, and the participants will be asked to perform as many repetitions as they can in 30s for each set. They will have 30 seconds to rest between sets (if they want more rest, we can let them more time but not exceed 60 seconds to limit the total amount of time for completing the exercise protocol) and 90 seconds to rest between exercises. Training sessions will occur twice per week with at least 24 hours between sessions. From the week 3rd of the intervention, the participants will perform the exercises with an adjustable weight vest with 5% of their body weight. In the middle intervention (post week 6 of the intervention which will be week 9 of the study), adolescents will be reevaluated for all the measures tested at the baseline. Weight vest will increase to 10% of their body weight for the last 4 weeks of the intervention.
  Arms: Loaded high intensity circuit training
Other: High intensity circuit training (HICT) — Participants will be familiarized to all the exercises. All exercises will have 3 sets, and the participants will be asked to perform as many repetitions as they can in 30s for each set. They will have 30 seconds to rest between sets (if they want more rest, we can let them more time but not exceed 60 seconds to limit the total amount of time for completing the exercise protocol) and 90 seconds to rest between exercises. Training sessions will occur twice per week with at least 24 hours between sessions.
  Arms: High Intensity Training

SUMMARY:
The purpose of this research study is to test the feasibility and response of a new exercise protocol on improving physical activity in adolescents with cerebral palsy.

DETAILED DESCRIPTION:
Only 25% of independent ambulatory children with spastic cerebral palsy (CP) meet the recommendations of time spent in physical activity (PA). Lack of PA during growing years is one of the root causes of obesity, diabetes, and hypertension. Children with CP are known to have poorer dynamic balance and weaker muscle strength than typically developing children, explaining their slower walking speeds, lower PA, and higher tripping and falling than typically developing children. These deficits markedly amplify in adolescence. Consequently, there is a critical need to mitigate deficits in muscle strength and dynamic balance in ambulatory adolescents with CP to increase PA. High intensity circuit training (HICT) vs progressive resistance training (PRT) improved PA to a greater degree in children with CP. Despite the use of HICT, PA in children with CP is still below the recommended level. Our new exercise protocol combines the principles of HICT and PRT in one training program to improve PA in adolescences with CP. The aim of this study is to test the feasibility and response of a new exercise protocol on improving physical activity in adolescents with cerebral palsy. In order to test the feasibility and response of the new exercise protocol, this study will have 3 groups of participants: 1) functionally loaded high intensity training exercise group, 2) a high intensity circuit training group, and 3) control group. For those two exercise groups, this study will include 4-week (weeks 2 - 5) exercise training program (including chair squat, side-step, split squat, heel raise, and jump). Children may/may not wear a weighted vest during exercising depend on their assigned group. For the non-exercise/control group, there is no intervention. Each group will have 2 sessions of baseline testing in week 1 and 1 session of post-testing in week 6. Coming for a single session of testing in week 9 is optional.

The following tests will be assessed before and after the exercise training program for all the groups: Lower limb strength and power via jump tests, balance via four-square step test, lateral step-up test, timed up and go tests, and walking tests. Their muscle and tendon stiffness will be assessed via a handheld device. Free living PA will be assessed via waist-worn accelerometers and questionnaires. Testing will be performed at 5 time points: tests at the first week (baseline 1 and baseline 2), sixth week (post training), ninth week (the follow up) of the study.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed diagnosis of spastic cerebral palsy or spina bifida
* independent ambulatory
* able to follow verbal instructions
* willing to commit to participate for the full study

Exclusion Criteria:

* had previous orthopedic surgery or botulinum toxin A injection in the lower limb within past 6 months
* had a structured lower limb exercise training within the past 6 months
* plan to go for any structured outside-of the-study exercise training
* had any heart, lung, vision, hearing or bodily issues that can interfere with participation and completion of the study
* had any other diseases that interfere with physical activity.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Week 1
  Step counts.
Physical Activity | Week 6
  Step counts. An increase in step counts is expected.

SECONDARY OUTCOMES:
Muscle Stiffness | Week 1
  Measure muscle and tendon stiffness. A decrease in stiffness is expected.
Muscle Stiffness | Week 6
  Measure muscle and tendon stiffness. A decrease in stiffness is expected.
Four square step test | Week 1
  Measure by time to complete test. A decrease in time completed is expected.
Four square step test | Week 6
  Measure by time to complete test. A decrease in time completed is expected.
Jumping test | Week 1
  Measure by jump height. An increase in jump height is expected.
Jumping test | Week 6
  Measure by jump height. An increase in jump height is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Harshvardhan Singh, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No